CLINICAL TRIAL: NCT04527263
Title: BUILDING UP A DIAGNOSTIC MODEL OF ACUTE APPENDICITIS IN CHILDREN USING URINARY 5-HYDROXY INDOL ACETIC ACID
Brief Title: Urinary 5-HIAA for Diagnosis of Acute Appendicitis in Children, Does it Help?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammad Gharieb Mohammad Khirallah, assistant professor of pediatric surgery, Tanta University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 33944/7/20
Record Dates: First submitted 2020-08-22; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Diagnosis of Acute Appendicitis in Children
Keywords: appendicitis, children, 5-HIAA, scoring systems
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): subjected to institutional protocol of diagnosis of acute appendicitis
  Interventions: Diagnostic Test: measurement of urinary 5-HIAA
- group B (Active Comparator): subjected to institutional protocol of diagnosis of acute appendicitis plus measurement of urinary 5-HIAA
  Interventions: Diagnostic Test: measurement of urinary 5-HIAA

INTERVENTIONS:
Diagnostic Test: measurement of urinary 5-HIAA — urinary assessment of 5-HIAA

SUMMARY:
it is randomized control study. two groups of children (n=191) were divided into two groups A and B. Group A included children subjected to the classical protocol of diagnosis of acute appendicitis. this protocol consisted of pediatric appendicitis score evaluation, pelvi abdominal ultrasound and measurement of serum CRP. Group B, children had the same previous assessment plus measurement of urinary 5-HIAA.

DETAILED DESCRIPTION:
1.1- Study design: Patients were randomly categorized into two groups A and B. Randomization was achieved using closed envelop method.

Group A (n= 95) included patients that were evaluated using our institutional protocol. This protocol consists of assessment of children using PAS, ultrasound of abdomen and pelvis and serum levels of C-reactive protein.

Group B (n= 96) included children that were evaluated by our institutional protocol. In addition, all children gave a mid- stream urine sample for spot urinary 5-HIAA detection. Detailed history was taken. This mainly was to exclude cases with history of foods or drugs that may affect level of serotonin in urine such as mono amino oxidase inhibitors.

All related clinical data and laboratory investigations were recorded. 1.2- Quantitation of urinary 5-HIAA level: From each participant, a random urine sample was obtained to assess the urinary 5-HIAA level using a solid phase competitive enzyme-linked immunosorbent assay (ELISA) technique. The commercial kit was purchased and provided by LDN, DN Labor Diagnosika Nord GmbH & Co. Nordhorn, Germany; Catalog #: BA E-1900. As stated by the manufacturer, the urine samples were methylated to derivatize the 5-HIAA. On the provided microtitre plate, the methylated standards, controls and samples are added. 5-HIAA antiserum was then added and incubated for 1 hour. After equilibration, excess free antigen and antigen-antibody complexes are washed out. The affixed bounded antibodies to the solid phase were detected by an anti-rabbit IgG-peroxidase conjugate using TMB as a substrate. The reaction is measured on a microplate reader (Tecan Spectra II, Switzerland), at 450 nm. Quantification of unknown sample concentration is processed by drawing a standard curve with known standard concentrations. The results of 5-HIAA were divided by urinary creatinine and expressed as mg/g creatinine. The inter-assay and intra-assay coefficient of variation were 10.8% and 8.6% respectively.

1.3- Clinical outcome: Diagnosis of acute appendicitis was confirmed by histopathological examination of resected appendix. According to operative findings and pathological reports, the condition ranged from negative appendix to different types of acute appendicitis (catarrhal, suppurative, perforated or gangrenous).

Children did not full filling the requirements for diagnosis as acute appendicitis were discharged on symptomatic treatment or after referral to pediatric emergency department.

Readmitted cases were recorded. 1.4- Statistical analysis: Statistical analysis was done using IBM SPSS V. 24 (IBM, NY, USA). A descriptive analysis was obtained for patients included in the study. Shapiro-Wilk test was conducted to check for normal distribution of dependent variables, such as urinary 5-HIAA, CRP and histopathological findings. X2 test was used to compare the categorical data. Student T-test was used to compare the normally distributed variable between two groups. Mann-Whitney U test and Kruskal-Wallis test were used for comparing the non-normally distributed variables of two and more than two groups, respectively. Binary logistic regression was performed to determine the independent predictors for acute appendicitis and to combine 5-HIAA and PAS results in both groups. Pearson correlation was used for correlating the urinary 5-HIAA with other acute appendicitis predictors. Receiver operating characteristic (ROC) curve was constructed to assess the diagnostic efficacy of acute appendicitis predictors. The optimal cutoff value for each predictor was assessed via the Youden index. The value of AUC ranged from 0.5 to 1.0. The ability of a diagnostic test to identify patients with appendicitis was considered optimal as AUC value reached closer to 1.0. P-value <0.05 was considered significant

ELIGIBILITY:
Inclusion Criteria:

* all children with suspected acute appendicitis

Exclusion Criteria:

* children received drugs that may affect normal values of urinary 5-HIAA as mono mono oxidase inhibitors

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 191 (Actual)
Dates: Start 2017-07-02 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
accurate diagnosis of acute appendicitis in children | 1 day
  number of cases that have been diagnosed as having acute appendicitis
decreasing incidence of negative appendectomy | 1 day
  number of cases that are not appendicitis and not operated
decreasing number of readmitted cases with diagnosis of acute appendicitis | 3 days
  number of cases that had been readmitted with diagnosis of acute appendicitis in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad G Mohammad, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided